CLINICAL TRIAL: NCT03260504
Title: A Phase I Trial of Interleukin-2 (Aldesleukin) and Pembrolizumab Combination Therapy for Patients With Advanced Renal Cell Carcinoma
Brief Title: Aldesleukin and Pembrolizumab in Treating Patients With Advanced or Metastatic Kidney Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: University of Washington (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Prometheus Laboratories (Industry)
Responsible Party: Principal Investigator, Scott Tykodi, MD, PhD, Associate Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9611; NCI-2017-01416 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RG1717068 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Advanced Clear Cell Renal Cell Carcinoma; Stage III Renal Cell Cancer; Stage IV Renal Cell Cancer; Metastatic Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Clear-cell metastatic renal cell carcinoma | interventions — aldesleukin; pembrolizumab; Immunoglobulin G

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, aldesleukin) (Experimental): Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Patients also receive aldesleukin subcutaneously (SC) 5 days per week for 6 weeks; or aldesleukin IV on days 2-6 of pembrolizumab cycles 1 and 2. Pembrolizumab treatment repeats every 3 weeks for 4 cycles per treatment course in the absence of clinical disease progression or unacceptable toxicity.
  Interventions: Biological: Aldesleukin; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Aldesleukin — Given SC or IV
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475; Immunoglobulin G4; Anti-(Human Programmed Cell Death 1)

SUMMARY:
This phase I trial studies the side effects and best dose of aldesleukin when given together with pembrolizumab in treating patients with kidney cancer that has spread to other parts of the body. Aldesleukin may stimulate white blood cells to kill kidney cancer cells. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to avoid recognition by immune cells. Giving aldesleukin and pembrolizumab may work better in treating patients with kidney cancer.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study of aldesleukin.

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Patients also receive aldesleukin subcutaneously (SC) 5 days per week for 6 weeks; or aldesleukin IV on days 2-6 of pembrolizumab cycles 1 and 2. Pembrolizumab treatment repeats every 3 weeks for 4 cycles per treatment course in the absence of clinical disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up via surveillance scans for every 3 months for up to 1 year or until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial
* Be >= 18 years of age on day of signing informed consent
* Have histologic confirmation of RCC with a clear cell component
* Have advanced (not amenable to potentially curative surgery) or metastatic RCC
* May have received previous systemic treatments or regimens for metastatic RCC. Prior therapy can include checkpoint blocking antibodies targeting PD-1, PD-L1, or cytotoxic Tlymphocyte-associated antigen-4 (CTLA-4) and/or targeted agents including TKIs, mTOR inhibitors, or bevacizumab. Patients may choose to receive study treatment as their initial therapy
* Previously treated patients must have documented disease progression after their last line of therapy
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Available tissue from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1,500 /mcL (within 14 days of treatment initiation)
* Platelets >= 100,000/mcL (within 14 days of treatment initiation)
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L (within 14 days of treatment initiation)
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or CrCl) >= 40 mL/min for subject with creatinine levels > 1.5 X institutional ULN; creatinine clearance should be calculated by Cockcroft-Gault (within 14 days of treatment initiation)
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (within 14 days of treatment initiation)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases (within 14 days of treatment initiation)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (dose level 2 and 3 patients only) (within 14 days of treatment initiation)
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (dose level 2 and 3 patients only) (within 14 days of treatment initiation)
* Forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) >= 65% of predicted (Testing performed prior to study screening are allowable. Pre-treatment testing must have been completed within 6 months of start of treatment) (within 14 days of treatment initiation)
* Left ventricular ejection fraction (LVEF) >= 50% measured by multigated acquisition (MUGA) scan, echo, or stress test study with myocardial perfusion imaging (Testing performed prior to study screening are allowable. Pre-treatment testing must have been completed within 6 months of start of treatment) (within 14 days of treatment initiation)
* Normal/negative cardiac stress testing with myocardial perfusion imaging OR cardiac catheterization with non-significant angiogram findings reviewed by a cardiology consultant (Testing performed prior to study screening are allowable. Pre-treatment testing must have been completed within 6 months of start of treatment) (within 14 days of treatment initiation)
* Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 140 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 200 days after the last dose of study therapy

Exclusion Criteria:

* Has received prior therapy with IL-2 or other investigational systemic cytokine therapy signaling through a common gamma-chain cytokine receptor including IL-7, IL-15 or IL-21
* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment
* Has had a prior monoclonal antibody within 4 weeks prior to study day I. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1
* Adverse events due to prior treatment must be resolved to < grade 1

  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* For patients previously treated with checkpoint blocking antibodies, no history of myocarditis, pneumonitis or nephritis of any grade associated with the prior treatment
* Has had autoimmune toxicity associated with prior checkpoint blocking antibodies requiring more than one drug class of immune suppressive therapy to resolve (e.g. steroid-refractory toxicity requiring infliximab, mycophenolate mofetil, tacrolimus or other immune suppressive agent) or requiring continuous immune suppression > 12 weeks, or having a severity judged to be life threatening by the investigator
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include locally curable cancers such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ of the cervix or breast that has undergone potentially curative therapy
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis

  * (Dose level 1) subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment
  * (Dose Level 2 and 3) subjects may not have any history of or current CNS metastases; baseline imaging of the brain is required within 28 days prior to the start of study treatments
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents; subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule; subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study; subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study
* Has history of (non-infectious) pneumonitis that required steroids or active, non-infectious pneumonitis
* Ongoing symptomatic cardiac dysrhythmias, uncontrolled atrial fibrillation, or prolongation of the corrected QT interval defined as > 450 msec for males and > 470 msec for female
* History of any of the following cardiovascular conditions within 6 months of enrollment: cardiac angioplasty or stenting, myocardial infarction, unstable angina, coronary artery bypass graft surgery, class III or IV congestive heart failure as defined by the New York Heart Association, symptomatic peripheral vascular disease, cerebrovascular accident, or transient ischemic attack
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days prior to the first dose of trial treatment; administration of killed vaccines are allowed; Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott S. Tykodi, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Period 1: Dose Level 1 (Pembrolizumab + SQ IL-2): Patients receive 200 mg pembrolizumab intravenously (IV) over 30 minutes on days 1, 22, 43, and 64.
  Patients also receive aldesleukin subcutaneously (SC) at 250,000 U/kg/dose, daily, 5 days/wk, week 1; 125,000 U/kg/dose, daily, 5 days/wk, weeks 2-6.
- Period 2: Dose Level 2 (Pembrolizumab + Low-Dose IV Bolus IL-2): Patients receive 200 mg pembrolizumab intravenously (IV) over 30 minutes on days 1, 22, 43, and 64.
  Patients also receive aldesleukin intravenously (IV) at 72,000 U/kg IV q 8 hrs x 14 doses days 2-6 (cycle 1); and days 23-27 (cycle 2) of a 12-week course.
Period: Overall Study
Arm/Group | Period 1: Dose Level 1 (Pembrolizumab + SQ IL-2) | Period 2: Dose Level 2 (Pembrolizumab + Low-Dose IV Bolus IL-2)
Started | 3 | 3
Completed | 3 | 2
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Period 1: Dose Level 1 (Pembrolizumab + SQ IL-2) | Period 2: Dose Level 2 (Pembrolizumab + Low-Dose IV Bolus IL-2) | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Median (Full Range); unit: Year] | 58 [57 to 67] | 59 [45 to 66] | 58 [45 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: The safety analysis was based on subjects who experienced toxicities as defined by CTCAE v5.0 criteria. Safety was assessed by quantifying the toxicities and laboratory abnormalities by grades experienced, including any serious adverse events (SAEs). Only treatment-related adverse events with an incidence rate of at least 2.5% are reported.
Time Frame: Adverse events were recorded from the time the consent form was signed through 30 days following the cessation of the study treatment for each participant. Each treatment course was 12 weeks and the maximum duration of treatment was 3 courses (36 weeks).
Measure: Number; unit: Adverse Events (CTCAE v5.0)
Arm/Group | Period 1: Dose Level 1 (Pembrolizumab + SQ IL-2) | Period 2: Dose Level 2 (Pembrolizumab + Low-Dose IV Bolus IL-2)
Number analyzed (Participants) | 3 | 3
Adverse Events (CTCAE v5.0) | 3 | 1

2. Secondary Outcome: Number of Participants With Objective Response
Description: Tumor imaging post-treatment compared to baseline imaging (MRI preferred or contrast CT); assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Best overall response rate (ORR) includes complete responders (CR): disappearance of all target lesions; and partial response (PR): at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Tumor imaging was collected at baseline after consent was obtained, every 12 weeks at end of a treatment course (max. 3 courses), and every 12 weeks after the cessation of study treatment for up to 1 year of surveillance follow-up for each participant.
Population: In Dose Level 2, one participant died before any staging assessment was collected and therefore could not be evaluated for objective response.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Dose Level 1 (Pembrolizumab + SQ IL-2) | Period 2: Dose Level 2 (Pembrolizumab + Low-Dose IV Bolus IL-2)
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

3. Secondary Outcome: Number of Participants With Objective Response or Stable Disease
Description: Tumor imaging post-treatment compared to baseline imaging (MRI preferred or contrast CT); assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Disease control rate includes CR; PR; stable disease: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (at least 20% in the sum of diameters of target lesions, taking as reference the smallest sum on study), taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: Dose Level 1 (Pembrolizumab + SQ IL-2) | Period 2: Dose Level 2 (Pembrolizumab + Low-Dose IV Bolus IL-2)
Number analyzed (Participants) | 3 | 2
Participants | 2 | 1

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival is defined from the time when the consent form was signed to when progressive disease was determined at tumor imaging assessment per protocol defined schedule or when death was reported.
Time Frame: as for outcome 2
Measure: Median (Full Range); unit: Months
Arm/Group | Period 1: Dose Level 1 (Pembrolizumab + SQ IL-2) | Period 2: Dose Level 2 (Pembrolizumab + Low-Dose IV Bolus IL-2)
Number analyzed (Participants) | 3 | 3
Months | 5.27 [2.33 to 5.40] | 2.67 [0.50 to 5.20]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time the consent form was signed through 30 days following the cessation of the study treatment for each participant. The maximum duration of treatment courses was 36 weeks. All-cause mortality was recorded from the time the consent form was signed for up to 1 year of surveillance following the end of study treatment for each participant.
Arm/Group | Period 1: Dose Level 1 (Pembrolizumab + SQ IL-2) | Period 2: Dose Level 2 (Pembrolizumab + Low-Dose IV Bolus IL-2)
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Dose Level 1 (Pembrolizumab + SQ IL-2) (N=3) | Period 2: Dose Level 2 (Pembrolizumab + Low-Dose IV Bolus IL-2) (N=3)
Myocarditis (Cardiac disorders) | 0 | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Dose Level 1 (Pembrolizumab + SQ IL-2) (N=3) | Period 2: Dose Level 2 (Pembrolizumab + Low-Dose IV Bolus IL-2) (N=3)
Generalized edema (General disorders) | 3 (7) | 3 (7)
Chills (General disorders) | 3 (6) | 3 (7)
Hypotension (Vascular disorders) | 1 (1) | 3 (12)
Nausea (Gastrointestinal disorders) | 3 (5) | 3 (6)
Creatinine increased (Investigations) | 2 (2) | 3 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (3)
Fever (General disorders) | 3 (4) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (5)
Headache (Nervous system disorders) | 2 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
Study enrollment was hampered by changes in frontline treatment options for advanced/metastatic RCC. There was a significant decrease of IL-2 therapy use at our cancer center starting in 2018 which coincided with the FDA approval of ICI-based regimens of nivolumab plus ipilimumab (2018), and pembrolizumab plus axitinib (2019). Study enrollment was also affected by the COVID-19 pandemic as our hospital prioritized efforts to inpatient care for patients with COVID-19 versus elective use of IL-2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT03260504/Prot_SAP_000.pdf